CLINICAL TRIAL: NCT00622960
Title: Comparison of High Monounsaturated Fat and High Carbohydrate Diets on Glycemic Control and Cardiovascular Risk Factors in Type 2 Diabetes
Brief Title: Effect of High Monounsaturated Fat Diet on Glycemic Control and Cardiovascular Risk Factors in Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Bonnie J. Brehm, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ADA 1-04-CR-05
Record Dates: First submitted 2008-02-13; First posted 2008-02-25 (Estimated); Last update posted 2008-02-25 (Estimated); Status verified 2008-02

CONDITIONS: Overweight; Obesity; Type 2 Diabetes
Keywords: obesity; type 2 diabetes; weight loss; monounsaturated fat; diet
MeSH Terms: conditions — Overweight; Obesity; Diabetes Mellitus, Type 2; Weight Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- High MUFA diet (Experimental): Those subjects assigned to a high monounsaturated fat diet
  Interventions: Other: High-MUFA diet
- High CHO diet (Active Comparator): Those subjects assigned to a high carbohydrate diet
  Interventions: Other: High-CHO diet

INTERVENTIONS:
Other: High-MUFA diet — The effects of high monounsaturated fat diet on body weight, body composition, lipid profile, and glycemic control.
  Arms: High MUFA diet
Other: High-CHO diet — The effects of high carbohydrate diet on body weight, body composition, lipid profile, and glycemic control.
  Arms: High CHO diet

SUMMARY:
The purpose of this proposed randomized, controlled trial is to compare the effects of high monounsaturated fat diets and high carbohydrate diets on body weight, body composition, glycemic control, plasma lipids, and other cardiovascular risk factors over a period of one year. At present, no such studies of free-living subjects have been performed. The specific aims of the proposed project are to test the hypotheses that (1) a high monounsaturated fat diet will produce greater weight loss/body fat loss and more successful weight maintenance than a high carbohydrate diet and (2) a high monounsaturated fat diet will result in an improved lipid profile and better glycemic control than a high carbohydrate diet.

DETAILED DESCRIPTION:
The incidence of type 2 diabetes has increased steadily over the last three decades. Although medical nutrition therapy is an integral component of diabetes management, nutrition recommendations for diabetes have often been based on clinical experience and expert consensus, rather than on carefully controlled clinical trials. The expert consensus on medical nutrition therapy is that carbohydrate and monounsaturated fat together should provide approximately 60-70% of total energy intake. This recommendation accommodates parties on both sides of a debate over what constitutes the optimal macronutrient composition of a diet for type 2 diabetic patients. On one side are proponents of high carbohydrate, low fat diets who contend that this regimen promotes the lowering of total- and LDL-cholesterol and is less calorically dense than diets containing a higher percentage of fat. On the other side are advocates of high monounsaturated fat, Mediterranean-type diets who cite data from short-term studies indicating that this approach decreases postprandial levels of plasma glucose, insulin, and triglycerides, and increases HDL-cholesterol more than isocaloric high carbohydrate diets. However, there is concern about the potential for high fat diets to increase energy intake and weight gain among free-living subjects. To make definitive, scientifically-based diet recommendations, it is essential that controlled long-term trials be conducted to demonstrate the health effects of specific percentages of monounsaturated fats and carbohydrates in the diets of persons with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* BMI of 27-40 kg/m2
* 30-75 years of age
* Stable body weight for the preceding 6 months
* Diagnosis of type 2 diabetes for at least 6 months prior to enrollment
* HbA1c of 6.5 to 9.0
* Treatment by diet or oral agents only

Exclusion Criteria:

* Pregnancy or lactation
* Active cardiac, pulmonary, renal, liver, or gastrointestinal disease
* Untreated thyroid disease or hypertension
* Hypertriglyceridemia with levels of TG > 500 mg/dl
* Use of insulin
* Use of specific medications that may alter lipid or glucose metabolism (other than the statins)
* Use of medications that commonly cause significant alterations in body weight (e.g., corticosteroids).

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2004-04; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
body weight | prior to and after 4, 8, and 12 months of dieting

SECONDARY OUTCOMES:
body fat | prior to and after 4, 8, and 12 months of dieting
blood pressure | prior to and after 4, 8, and 12 months of dieting
blood lipid profile | prior to and after 4, 8, and 12 months of dieting
glycemic control (glucose, insulin, and HbA1c) | prior to and after 4, 8, and 12 months of dieting

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie J Brehm, PhD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Brehm BJ, Lattin BL, Summer SS, Boback JA, Gilchrist GM, Jandacek RJ, D'Alessio DA. One-year comparison of a high-monounsaturated fat diet with a high-carbohydrate diet in type 2 diabetes. Diabetes Care. 2009 Feb;32(2):215-20. doi: 10.2337/dc08-0687. Epub 2008 Oct 28. PMID 18957534